CLINICAL TRIAL: NCT04398043
Title: Searching for SARS-CoV 2 in Personal Protective Equipment in Physicians in a University Hospital
Brief Title: SARS-CoV 2 in Personal Protective Equipment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas José de San Martín (Other)
Collaborators: Claudio Yaryour (Unknown); Fermepin Marcelo (Unknown); Luis Sarotto (Unknown); Federico Rodriguez Cairoli (Unknown); Angela Famiglieti (Unknown); Francisco Appiani (Unknown); Lucía Gallo Vaulet (Unknown)
Responsible Party: Principal Investigator, Bernardo Bergroth, MD, Chief of medical informatics, Hospital de Clinicas José de San Martín
Other Study IDs: rt PCR en EPP
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: rt PCR; COVID; Personal Protective Equipment PPE; SARS-CoV 2; Health Personnel Attitude; Virus Diseases
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The viral RNA of the sample will be purified using a commercial kit according to the manufacturer's instructions. Detection of SARS-CoV-2 will be performed on the viral RNA obtained from these samples by real-time RT-PCR according to the protocol of the US Center for Disease Control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SARS-CoV-2 transmission is frequently occurring in hospital settings, with numerous reported cases of nosocomial transmission highlighting the vulnerability of healthcare workers.

If products proved to be efficacious against COVID-19, why are so many HCW getting COVID-19? Is it related to experience? Is it generated by the exhaustive job? Is there any degree of relationship to stress? These questions are still without fully correct answers. Achieving global benefits for HCW is still waiting.

DETAILED DESCRIPTION:
Objective: To assess the extent of surface contamination PPE doctors (personal protective equipment) with SARS-CoV-2, immediately after evaluating ill patients.

COVID-19 is a recently emerging disease, in which much scientific information is being generated, but in which there are few certainties. This is due to work of poor methodological quality, but also due to the fact that it is a recent infection, which has only been developing for a few months. Given that most cases of infection in health personnel in the workplace come from contamination with personal protective equipment, it is necessary to determine there is any degree of contamination of PPE by the virus, as the critical areas where it can be located in the PPE as well. That is why this investigation, when trying to determine the location and degree of contamination of PPE by COVID-19, will allow the implementation of exhaustive care that leads to greater care for health personnel.

Target population: patients with a diagnosis of COVID-19 in patients admitted to a service in the General Ward and Intensive Care Unit or Coronary Unit of a University Hospital of C.A.B.A- (Argentina) Accessible population of adults patients with a diagnosis of COVID-19 admitted to the CN / Intensive Care Unit / Coronary Unit, while the research is in progress.

Population Definition Criteria: PPE of medical personnel in contact with hospitalized patients with SARS-CoV-2 positive swab, hospitalized in CM / UTI / UC wards.

Inclusion Criteria: Samples of personal protective equipment of health personnel who have been in contact with patients with positive viral RNA results in RT-real time PCR (rtPCR +) test for SARS-CoV-2 will be used.

Exclusion criteria:

PPE of health personnel who have been in contact with patients without confirmation of COVID-19 diagnosis.

Elimination Criteria: those patients who change the result of the positive viral load to negative viral load.

Time-space coordinates:

The research will be carried out from May 15, 2020 and will be carried out in the CM / UTI / UC rooms of the Hospital de Clínicas José de San Martín, in those patients with confirmed pathology of COVID-19 until reaching the necessary number of 16 patients.

2.2. Ethical objections to the project. This project is carried out under the ethical standards that govern human research in accordance with the National Law on Protection of Personal Data No. 25,326 (Habeas Data Law) and the Declaration of Helsinki in its latest version (Fortaleza 2013). The Bioethics and Teaching and Research Committee of the José de San Martín Clinic Hospital have given their approval to carry out the study.

ELIGIBILITY:
Inclusion Criteria:

* in patient with rtPCT possitive for SARSCoV-2 (interned in an intensive care unit, medical clinic room and coronary unit)

Exclusion Criteria:

* in pattient with negattive rtPCT for SARSCoV-2

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In patients in a University Hospital with COVID 19 desease
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Asses surface contamination personel protective equipment | 2 months
  To assess the prevalence of surface contamination with COVID-19 from personal protective equipment (PPE) worn by medical doctors, immediately after evaluating sick patients

SECONDARY OUTCOMES:
Virus charge cuantification | 2 months
  Quantify the amount of COVID-19 in the PPE doctor´s in contact with infected patients.
Place in PPE contamination | 2 month
  Determine the most frequent location of viruses inPPE

OTHER OUTCOMES:
Prevention risk advice | 2 month
  using the information found, carry out tips to reduce the risk of contagion

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Yaryour, MD, Study Chair — Hospital de Clínicas José de San Martín, UBA

IPD SHARING:
Plan to Share IPD: Undecided
It depnds on formulations

REFERENCES:
- [Background] The Lancet. COVID-19: protecting health-care workers. Lancet. 2020 Mar 21;395(10228):922. doi: 10.1016/S0140-6736(20)30644-9. No abstract available. PMID 32199474
- [Background] Morawska L, Cao J. Airborne transmission of SARS-CoV-2: The world should face the reality. Environ Int. 2020 Jun;139:105730. doi: 10.1016/j.envint.2020.105730. Epub 2020 Apr 10. PMID 32294574
- [Background] Meselson M. Droplets and Aerosols in the Transmission of SARS-CoV-2. N Engl J Med. 2020 May 21;382(21):2063. doi: 10.1056/NEJMc2009324. Epub 2020 Apr 15. No abstract available. PMID 32294374
- [Background] Assessment of N95 respirator decontamination and re-use for SARS-CoV-2 Robert Fischer, View ORCID ProfileDylan H Morris, Neeltje van Doremalen, Shanda Sarchette, Jeremiah Matson, Trenton Bushmaker, Claude Kwe Yinda, Stephanie Seifert, Amandine Gamble, Brandi Williamson, Seth Judson, Emmie de Wit, Jamie Lloyd-Smith, View ORCID ProfileVincent Munster doi: https://doi.org/10.1101/2020.04.11.20062018
- [Background] Loeffelholz MJ, Tang YW. Laboratory diagnosis of emerging human coronavirus infections - the state of the art. Emerg Microbes Infect. 2020 Dec;9(1):747-756. doi: 10.1080/22221751.2020.1745095. PMID 32196430
- [Background] Maguire BJ, Guerin PJ. A living systematic review protocol for COVID-19 clinical trial registrations. Wellcome Open Res. 2020 Apr 2;5:60. doi: 10.12688/wellcomeopenres.15821.1. eCollection 2020. PMID 32292826